CLINICAL TRIAL: NCT05946317
Title: Evaluation of Sir William Kelsey Fry Technique in Lingual Surgical Removal of Impacted Lower Third Molar With Retraction Lingual Nerve
Brief Title: Removal of Impacted Molars With Lingual Split Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TishreenU - Maxillofacial surg
Record Dates: First submitted 2023-06-12; First posted 2023-07-14 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Lingual Nerve Injuries
Keywords: Impacted third molar; lingual nerve; lingual flap retractor
MeSH Terms: conditions — Lingual Nerve Injuries

STUDY DESIGN:
Intervention Model Description: The research sample included 20 patients from the Faculty of Dentistry in Tishreen University and maxillofacial surgery department in Tishreen Hospital who had have an impacted mandibular third molar indicated for extraction and their age under 25 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lingual nerve function assessed after removal of Impacted mandibular third molar (Experimental): 20 patients who had have an impacted mandibular third molar indicated for extraction by lingual split technique with using Walter's lingual retractor for retracting lingual flap.
  The neurological function of the lingual nerve was assessed after the demise of local anesthesia, then the location of the disorder and taste function and healing time are determined by sensory neurological tests on a graphic map that divides the tongue into sextants.
  Interventions: Procedure: Lingual nerve function assessed after removal of mandibular third molar with lingual split technique

INTERVENTIONS:
Procedure: Lingual nerve function assessed after removal of mandibular third molar with lingual split technique — The lingual split technique is based on using chisel and hammer in bone removing. After the buccal and lingual flaps are raised and retracted. Two buccal bone cutting with horizontal cutting up between them are performed, The disto-lingual bone fragment is fractured inward by placing the cutting edge of the chisel at 45 degrees with the surface of the bone and directed towards the lower second premolar of the opposite side. By maintaining the cutting edge of the chisel parallel to the external oblique ridge, a few light taps with the mallet will separate the lingual plate from the rest of the alveolar bone. And it released from soft tissues, buccally force is applied to roll the whole tooth lingually. The neurological function of the lingual nerve was assessed after the demise of local anesthesia, then the location of the disorder and taste function and healing time are determined by sensory neurological tests on a graphic map that divides the tongue into sextants.

SUMMARY:
This research assesses removal of mandibular third molars by the lingual split technique with using Walter's lingual retractor for retracting lingual flap, and evaluates the lingual nerve injury that may result after applying this technique. The research sample included 20 patients and their age under 25 years where the grain is clear. The lingual nerve is assessed by sensory neurological tests on a graphic map that divides the tongue into sextants.

DETAILED DESCRIPTION:
Although the scope of oral and maxillofacial surgery has expanded in many directions recently, the common or recurrent practice remains dentoalveolar surgery including impaction surgery. The main indication to extract is whether the third molar has involved in a disease process.

Permanent injury of lingual and chorda tympani nerve (influenced by taste sensations) following removal mandibular third molar remains a clinical problem in oral and maxillofacial surgery. To reduce the risk of lingual nerve injury, the current protocols in North America accentuate raising a buccal flap and following a buccal approach during removal impacted mandibular third molar. However, there was no uniform success as a clinical reality showed. Many patients are still being referred to specialist centers for the management of lingual nerve injury. In most cases, the surgeon was not discerned of any incident that could cause the neurological injury. The alternative technique is Lingual split technique.

Lingual split technique for removal impacted mandibular third molars introduced by Kelsey Fry and described by Ward in 1956 by removing a thin piece of disto-lingual bone and removing the tooth lingually. This technique is initially designed to remove distal and lingually inclined impacted mandibular third molar. This technique has not received much appreciation because of potential associated morbidity. Complications with this technique are potential damage to the lingual nerve, increasing hemorrhage from the lingual cohesive soft tissue, infection expansion to the sublingual or sublingual spaces and edema close to the airway. Several modifications have been made on the lingual split technique which they have reduced trauma and prevent complications. The advantages of this technique are easy, safety, less time-consuming and minimal tissue trauma and complications with good outcomes. Also, it allows obtaining the impacted third molar in one piece, and may be used as a donor tooth for non-restorable molar replacement. It has the advantage of reducing the volume of residual thrombosis when using sauzerization means. Few studies look specifically at the lingual split technique, which has been criticized for causing a high rate of lingual nerve injury and excluded for centuries.

The independent basis in lingual spilt technique is that the lingual plate is much thinner than the buccal, especially in cases where the tooth is fully bone impacting. It is suitable for use in young patients only with a flexible bone where the grain is clear.6 The direction of the grain and the presence of the lingual prominence of the alveolar process allow the desired part of the bone plate to easily detach by chiseling and this makes the technique more rapid.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have impacted mandibular third molar indicated for removal.
* Patients are healthy and have no systemic diseases (ASA1 ASA2).
* Patient's age is less than 25 years where the bone grain is still present and the use of the chisel and hammer is permitted.
* Patient's consent to surgical work and inclusion in the research.

Exclusion Criteria:

* A deep impacted mandibular third molar which is close proximately to the neuro-vascular package, deep horizontal impaction, extreme disto-angular impaction.
* Patient's age is over 25 years.
* The lingual plate is thick.

Ages: 19 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
Lingual nerve injury location | 6 hours after the surgical procedure of removal of impacted mandibular third molar.
  The location of the disorder on the tongue is determined on a graphic map that divides the tongue into six sextants in each side: middle apical, lateral apical, middle, lateral, middle posterior and lateral posterior.
Nerve discrepancy | 6 hours after the surgical procedure of removal of impacted mandibular third molar.
  0 : No sensational impairment
  1. : Mild loss of sensation
  2. : Moderate loss of sensation
  3. : Severe loss of sensation
Taste function | 6 hours after the surgical procedure of removal of impacted mandibular third molar.
  Taste function is assessed by Taste sensation tests of sweetness, saltiness, acidity and bitterness.

SECONDARY OUTCOMES:
Healing time | Two weeks after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.
Healing time | Four weeks after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.
Healing time | Six weeks after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.
Healing time | Two months after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.
Healing time | Four months after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.
Healing time | Six months after the surgical procedure.
  The McGill Pain Questionnaire (MPQ), it is a useful tool for monitoring progression of neurosensory recovery. This is a 10 cm five-degree scale, with a degree marked every 2.5 cm.
  1. : complete absence of sensation.
  2. : Almost no sensation.
  3. : Reduced sensation.
  4. : Almost normal sensation.
  5. : Fully normal sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Karim Khalil, PHD, Study Chair — Tishreen University; Alaa Alaji, Master, Principal Investigator — Tishreen University
Locations (1):
- Alaa Alaji, Latakia, Syria

REFERENCES:
- [Background] Rud J. Reevaluation of the lingual split-bone technique for removal of impacted mandibular third molars. J Oral Maxillofac Surg. 1984 Feb;42(2):114-7. doi: 10.1016/0278-2391(84)90323-9. No abstract available. PMID 6582236
- [Background] Farish SE, Bouloux GF. General technique of third molar removal. Oral Maxillofac Surg Clin North Am. 2007 Feb;19(1):23-43, v-vi. doi: 10.1016/j.coms.2006.11.012. PMID 18088862
- [Background] Pippi R, Spota A, Santoro M. Prevention of Lingual Nerve Injury in Third Molar Surgery: Literature Review. J Oral Maxillofac Surg. 2017 May;75(5):890-900. doi: 10.1016/j.joms.2016.12.040. Epub 2017 Jan 4. PMID 28142010
- [Background] Pogrel MA, Goldman KE. Lingual flap retraction for third molar removal. J Oral Maxillofac Surg. 2004 Sep;62(9):1125-30. doi: 10.1016/j.joms.2004.04.013. PMID 15346365
- [Background] Steel B. Lingual split versus surgical bur technique in the extraction of impacted mandibular third molars: a systematic review. Oral Surg Oral Med Oral Pathol Oral Radiol. 2012 Sep;114(3):294-302. doi: 10.1016/j.tripleo.2011.07.028. Epub 2012 Jan 27. PMID 22883979
- [Background] Smith MH, Lung KE. Nerve injuries after dental injection: a review of the literature. J Can Dent Assoc. 2006 Jul-Aug;72(6):559-64. PMID 16884649